CLINICAL TRIAL: NCT01695395
Title: Mental Health Care Provision for Adults With Mental Retardation and a Psychiatric Diagnosis
Brief Title: Mental Health Care Provision for Adults With Intellectual Disability and a Mental Disorder
Acronym: MEMENTA
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Dr. Matthias Schützwohl, PD, Technische Universität Dresden
Other Study IDs: BMBF-01GY1134
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Mental Disorder; Intellectual Disability
Keywords: intellectual disability; mental disorder; dual diagnosis; provision; needs assessment; quality of life
MeSH Terms: conditions — Mental Disorders; Intellectual Disability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Intellectual disabled adults without a mental disorder
- Intellectual disabled adults with a mental disorder

SUMMARY:
Quality of mental health services provision for adults with intellectual disability and comorbid mental disorder is considered inadequate and therefore in need of further improvement. However, empirical findings on this topic are rather scarce. The MEMENTA-study therefore aims to compare mild and moderate intellectual disabled adults with a comorbid mental disorder to mild and moderate intellectual disabled adults who do not have a comorbid mental disorder with respect to clinical parameters. The MEMENTA-study is an observational, epidemiological, cross-sectional study. A representative sample of the target population is realised by the assessment of approximately n=600 intellectual disabled adults working at specialized facilities (sheltered workshops). A cluster sampling with probability proportional to institution and size (n of overall employed persons) will be followed by a simple random sampling of persons of these clustered facilities. A number of parameters such as severity of mental health impairment, needs for care, quality of life (QoL), caregiver burden, health services utilization, and costs for care will be assessed by using a set of well-established standardised instruments. Quality of mental health care will be assessed and examined by open questions to intellectual disabled adults with a comorbid mental disorder as well as informal caregivers and staff of caring institutions.

ELIGIBILITY:
Inclusion Criteria:

* mild or moderate intellectual disability
* adults aged between 18-65 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are adults with mild or moderate intellectual disability.
Sampling Method: Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2012-02; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Mental Health status | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Schützwohl, PD Dr., Principal Investigator — TU Dresden
Locations (3):
- Germany (3):
  - Psychiatric Health Service Research Group, Department of Psychiatry and Psychotherapy, Carl Gustav Carus University Hospital, Dresden, Saxony
  - Central Institute of Mental Health, Mannheim
  - Mental Health Services RU, Department of Psychiatry II, Ulm University, Ulm

REFERENCES:
- [Derived] Koch A, Vogel A, Holzmann M, Pfennig A, Salize HJ, Puschner B, Schutzwohl M. MEMENTA-'Mental healthcare provision for adults with intellectual disability and a mental disorder'. A cross-sectional epidemiological multisite study assessing prevalence of psychiatric symptomatology, needs for care and quality of healthcare provision for adults with intellectual disability in Germany: a study protocol. BMJ Open. 2014 May 20;4(5):e004878. doi: 10.1136/bmjopen-2014-004878. PMID 24844270